CLINICAL TRIAL: NCT05373862
Title: Clinical Evaluation of Arrhythmia Mapping With a Globe-Shaped, High-Density, Multi-Electrode Mapping Catheter
Brief Title: A Study Assessing Arrhythmia Mapping With a Globe-Shaped, High-Density, Multi-Electrode Mapping Catheter
Acronym: COSMOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BWI_2021_01; CIV-22-03-039047 (Other: EUDAMED CIV-ID); BWI_2021_01 (Other: Biosense Webster, Inc.)
Record Dates: First submitted 2022-05-10; First posted 2022-05-13 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Scar-related Atrial Tachycardia; Persistent Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Ventricular Tachycardia; Premature Ventricular Complex
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia, Ventricular; Ventricular Premature Complexes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Globe-Shaped, High-Density, Multi-Electrode Mapping Catheter (Experimental): Participants with cardiac arrhythmias/ablation history who are scheduled to have a clinically-indicated catheter mapping and ablation procedure of arrhythmia management for atrial and ventricular procedures will be using multi-electrode mapping catheter.
  Interventions: Device: Globe-Shaped, High-Density, Multi-Electrode Mapping Catheter

INTERVENTIONS:
Device: Globe-Shaped, High-Density, Multi-Electrode Mapping Catheter — Participants scheduled to have a clinically-indicated catheter mapping and ablation procedure using globe-shaped, high-density, multi-electrode mapping catheter for management of atrial procedure (scar-related atrial tachycardia, persistent atrial fibrillation, paroxysmal atrial fibrillation) and Ventricular procedures (ventricular tachycardia, premature ventricular complex).

SUMMARY:
The purpose of this study is to assess the performance and safety for the use of the investigational catheter for intracardiac mapping in the atria and ventricles.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with and candidate for clinically-indicated catheter mapping and ablation procedure for the management of ventricular tachycardia, premature ventricular complex, atrial tachycardia or atrial fibrillation (participants having undergone a previous ablation procedure may be included)
* At least one episode of the targeted arrhythmia (ventricular tachycardia, premature ventricular complex, atrial tachycardia or atrial fibrillation) must have been documented by electrocardiogram (ECG), Holter, loop recorder, telemetry, implanted device, or transtelephonic monitoring within 12 months of enrollment
* Signed participants Informed Consent Form (ICF)
* Able and willing to comply with all pre-, post-, and follow-up testing and requirements

Exclusion Criteria:

* Diagnosed with an arrhythmia requiring epicardial mapping
* Study arrhythmia secondary to reversible cause, or secondary to electrolyte imbalance, thyroid disease, or non-cardiac cause
* Atrial arrhythmias: participants with a left atrial size greater than (>) 55 millimeters (mm)
* Left Ventricular Ejection Fraction (LVEF) less than or equal to (<=) 25 percent (%) for participants with ventricular arrhythmia
* LVEF <= 40% for participants with atrial arrhythmia
* Documented intracardiac thrombus as detected on imaging within 24 hours prior to insertion of the investigational catheter
* Contraindication to anticoagulation (that is heparin, warfarin, dabigatran)
* History of blood clotting or bleeding abnormalities (example, hypercoagulable state)
* Myocardial infarction within the past 2 months (60 days)
* Documented thromboembolic event (including Transient Ischemic Attack [TIA]) within the past 12 months (365 days)
* Uncontrolled heart failure or New York Heart Association (NYHA) function class IV
* Implanted with a pacemaker or intracardiac cardiac defibrillator within the past 6 weeks (42 days)
* Participants with known untreatable allergy to contrast media
* Active illness or active systemic infection or sepsis
* Diagnosed atrial or ventricular myxoma, interatrial baffle or patch, tumor or other abnormality that precludes catheter introduction or manipulation
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study
* Participants that have ever undergone a percutaneous or surgical valvular cardiac procedure (that is, ventriculotomy, atriotomy, and valve repair or replacement and presence of a prosthetic valve)
* Any cardiac surgery within the past 60 days (2 months) (includes Percutaneous Coronary Intervention [PCI])
* Atrial septal closure within the past 6 weeks (42 days)
* Presence of a condition that precludes vascular access
* Women who are pregnant (as evidenced by pregnancy test if pre-menopausal), lactating, or who are of childbearing age and plan on becoming pregnant during the course of the clinical investigation
* Categorized as vulnerable population and requires special treatment with respect to safeguards of well-being
* Concurrent enrollment in an investigational study evaluating another device or drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biosense Webster, Inc. Clinical Trial, Study Director — Biosense Webster, Inc.
Locations (4):
- Belgium (2):
  - Onze-Lieve-Vrouw (OLV) Ziekenhuis, Aalst
  - Universitair Ziekenhuis (UZ) Brussel, Brussels
- University Hospital Center Split, Split, Croatia
- Ospedale Generale Regionale Francesco Miulli (F. Miulli), Acquaviva delle Fonti, Italy

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Bick RL, Frenkel EP. Clinical aspects of heparin-induced thrombocytopenia and thrombosis and other side effects of heparin therapy. Clin Appl Thromb Hemost. 1999 Oct;5 Suppl 1:S7-15. doi: 10.1177/10760296990050s103. PMID 10726030
- [Background] Cox B, Durieux ME, Marcus MA. Toxicity of local anaesthetics. Best Pract Res Clin Anaesthesiol. 2003 Mar;17(1):111-36. doi: 10.1053/bean.2003.0275. PMID 12751552
- [Background] Gruchalla RS. 10. Drug allergy. J Allergy Clin Immunol. 2003 Feb;111(2 Suppl):S548-59. doi: 10.1067/mai.2003.93. PMID 12592301
- [Background] Mertes PM, Laxenaire MC. Allergic reactions occurring during anaesthesia. Eur J Anaesthesiol. 2002 Apr;19(4):240-62. doi: 10.1017/s0265021502000418. PMID 12074414
- [Background] Morcos SK, Thomsen HS, Webb JA; Contrast Media Safety Committee of the European Society of Urogenital Radiology. Prevention of generalized reactions to contrast media: a consensus report and guidelines. Eur Radiol. 2001;11(9):1720-8. doi: 10.1007/s003300000778. PMID 11511894
- [Background] Lin, A.C. and D.J. Wilber, Complications Associated With Radiofrequency Catheter Ablation, in Radiofrequency catheter ablation of cardiac arrhythmias: basic concepts and clinical applications, S.K. Huang and D.J. Wilber, Editors. 2000, Futura: Armonk, N.Y. p. 737-746.
- [Background] Scheinman MM, Huang S. The 1998 NASPE prospective catheter ablation registry. Pacing Clin Electrophysiol. 2000 Jun;23(6):1020-8. doi: 10.1111/j.1540-8159.2000.tb00891.x. PMID 10879389
- [Background] Mar PL, Chong L, Perez A, Lakkireddy D, Gopinathannair R. Entrapment of diagnostic catheter within Advisor HD grid mapping catheter. J Cardiovasc Electrophysiol. 2021 Mar;32(3):860-861. doi: 10.1111/jce.14893. Epub 2021 Jan 28. PMID 33476457
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation: Executive summary. J Arrhythm. 2017 Oct;33(5):369-409. doi: 10.1016/j.joa.2017.08.001. Epub 2017 Sep 15. No abstract available. PMID 29021841
- [Background] Cappato R, Calkins H, Chen SA, Davies W, Iesaka Y, Kalman J, Kim YH, Klein G, Natale A, Packer D, Skanes A, Ambrogi F, Biganzoli E. Updated worldwide survey on the methods, efficacy, and safety of catheter ablation for human atrial fibrillation. Circ Arrhythm Electrophysiol. 2010 Feb;3(1):32-8. doi: 10.1161/CIRCEP.109.859116. Epub 2009 Dec 7. PMID 19995881
- [Background] Gerstenfeld EP, Guerra P, Sparks PB, Hattori K, Lesh MD. Clinical outcome after radiofrequency catheter ablation of focal atrial fibrillation triggers. J Cardiovasc Electrophysiol. 2001 Aug;12(8):900-8. doi: 10.1046/j.1540-8167.2001.00900.x. PMID 11513440
- [Background] Kovoor P, Ricciardello M, Collins L, Uther JB, Ross DL. Risk to patients from radiation associated with radiofrequency ablation for supraventricular tachycardia. Circulation. 1998 Oct 13;98(15):1534-40. doi: 10.1161/01.cir.98.15.1534. PMID 9769307
- [Background] Nahass GT. Fluoroscopy and the skin: implications for radiofrequency catheter ablation. Am J Cardiol. 1995 Jul 15;76(3):174-6. doi: 10.1016/s0002-9149(99)80053-8. No abstract available. PMID 7611155
- [Background] Calkins H, Niklason L, Sousa J, el-Atassi R, Langberg J, Morady F. Radiation exposure during radiofrequency catheter ablation of accessory atrioventricular connections. Circulation. 1991 Dec;84(6):2376-82. doi: 10.1161/01.cir.84.6.2376. PMID 1959193
- [Background] Cronin EM, Bogun FM, Maury P, Peichl P, Chen M, Namboodiri N, Aguinaga L, Leite LR, Al-Khatib SM, Anter E, Berruezo A, Callans DJ, Chung MK, Cuculich P, d'Avila A, Deal BJ, Della Bella P, Deneke T, Dickfeld TM, Hadid C, Haqqani HM, Kay GN, Latchamsetty R, Marchlinski F, Miller JM, Nogami A, Patel AR, Pathak RK, Saenz Morales LC, Santangeli P, Sapp JL, Sarkozy A, Soejima K, Stevenson WG, Tedrow UB, Tzou WS, Varma N, Zeppenfeld K; ESC Scientific Document Group. 2019 HRS/EHRA/APHRS/LAHRS expert consensus statement on catheter ablation of ventricular arrhythmias. Europace. 2019 Aug 1;21(8):1143-1144. doi: 10.1093/europace/euz132. PMID 31075787
- [Background] Raymond JM, Sacher F, Winslow R, Tedrow U, Stevenson WG. Catheter ablation for scar-related ventricular tachycardias. Curr Probl Cardiol. 2009 May;34(5):225-70. doi: 10.1016/j.cpcardiol.2009.01.002. PMID 19348944

RESULTS

PARTICIPANT FLOW:
Groups:
- Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter): Participants diagnosed with cardiac arrhythmias who were scheduled to have a clinically-indicated catheter mapping and ablation procedure of arrhythmia management for atrial and ventricular procedures, underwent pre-ablation mapping of the chambers of interest using the multi-electrode ECG mapping catheter (investigational catheter) prior to a standard of care ablation procedure.
Period: Overall Study
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (15.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pre-ablation Mapping Requirements and Clinically Indicated Mapping Performed With the Investigational Catheter Without Resort to Non-study Mapping Catheter(s)
Description: Number of participants with pre-ablation mapping requirements and clinically indicated mapping performed with the investigational catheter without resort to non-study mapping catheter(s) were reported.
Time Frame: Up to 7 days of index procedure on Day 1
Population: Per-protocol analysis set included all participants who completed the protocol-required "pre-ablation mapping" with the investigational catheter.
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
Number analyzed (Participants) | 40
Participants | 40

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) Within 7 Days of Index Procedure Related to the Investigational Catheter
Description: Number of participants with SAEs within 7 days of index procedure related to the investigational catheter were reported. An adverse event (AE) is any untoward medical occurrence in a participant whether or not related to the investigational device. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to 7 days of index procedure on Day 1
Population: The safety analysis set consisted of all enrolled participants who underwent insertion of the study catheter.
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
Number analyzed (Participants) | 40
Participants | 1

3. Secondary Outcome: Number of Responders for Physician Assessment for Maneuverability and Handling
Description: Number of responders for physician assessment for maneuverability & handling were reported. A post-procedure survey of 11 questions, each with individual sub-questions were asked. Each question/sub-question was answered by the physician using a Likert scale of 1 to 7 (1=poor and 7=excellent). Responders refers to participants with physician assessment for maneuverability and handling.
Time Frame: Up to 29 weeks
Population: The safety analysis set consisted of all enrolled participants who underwent insertion of the study catheter. Here, 'n' (number analyzed) is defined as participants analyzed for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
Number analyzed (Participants) | 40
Participants
  Ability to Deploy (Left Atrium): Score 1: number analyzed (Participants) | 32
  Ability to Deploy (Left Atrium): Score 1 | 0
  Ability to Deploy (Left Atrium): Score 2: number analyzed (Participants) | 32
  Ability to Deploy (Left Atrium): Score 2 | 1
  Ability to Deploy (Left Atrium): Score 3: number analyzed (Participants) | 32
  Ability to Deploy (Left Atrium): Score 3 | 1
  Ability to Deploy (Left Atrium): Score 4: number analyzed (Participants) | 32
  Ability to Deploy (Left Atrium): Score 4 | 6
  Ability to Deploy (Left Atrium): Score 5: number analyzed (Participants) | 32
  Ability to Deploy (Left Atrium): Score 5 | 7
  Ability to Deploy (Left Atrium): Score 6: number analyzed (Participants) | 32
  Ability to Deploy (Left Atrium): Score 6 | 14
  Ability to Deploy (Left Atrium): Score 7: number analyzed (Participants) | 32
  Ability to Deploy (Left Atrium): Score 7 | 3
  Ability to Deploy (Right Atrium): Score 1: number analyzed (Participants) | 20
  Ability to Deploy (Right Atrium): Score 1 | 0
  Ability to Deploy (Right Atrium): Score 2: number analyzed (Participants) | 20
  Ability to Deploy (Right Atrium): Score 2 | 0
  Ability to Deploy (Right Atrium): Score 3: number analyzed (Participants) | 20
  Ability to Deploy (Right Atrium): Score 3 | 1
  Ability to Deploy (Right Atrium): Score 4: number analyzed (Participants) | 20
  Ability to Deploy (Right Atrium): Score 4 | 4
  Ability to Deploy (Right Atrium): Score 5: number analyzed (Participants) | 20
  Ability to Deploy (Right Atrium): Score 5 | 4
  Ability to Deploy (Right Atrium): Score 6: number analyzed (Participants) | 20
  Ability to Deploy (Right Atrium): Score 6 | 9
  Ability to Deploy (Right Atrium): Score 7: number analyzed (Participants) | 20
  Ability to Deploy (Right Atrium): Score 7 | 2
  Ability to Deploy (Left Ventricle): Score 1: number analyzed (Participants) | 2
  Ability to Deploy (Left Ventricle): Score 1 | 0
  Ability to Deploy (Left Ventricle): Score 2: number analyzed (Participants) | 2
  Ability to Deploy (Left Ventricle): Score 2 | 0
  Ability to Deploy (Left Ventricle): Score 3: number analyzed (Participants) | 2
  Ability to Deploy (Left Ventricle): Score 3 | 0
  Ability to Deploy (Left Ventricle): Score 4: number analyzed (Participants) | 2
  Ability to Deploy (Left Ventricle): Score 4 | 0
  Ability to Deploy (Left Ventricle): Score 5: number analyzed (Participants) | 2
  Ability to Deploy (Left Ventricle): Score 5 | 0
  Ability to Deploy (Left Ventricle): Score 6: number analyzed (Participants) | 2
  Ability to Deploy (Left Ventricle): Score 6 | 1
  Ability to Deploy (Left Ventricle): Score 7: number analyzed (Participants) | 2
  Ability to Deploy (Left Ventricle): Score 7 | 1
  Ability to Deploy (Right Ventricle): Score 1: number analyzed (Participants) | 8
  Ability to Deploy (Right Ventricle): Score 1 | 0
  Ability to Deploy (Right Ventricle): Score 2: number analyzed (Participants) | 8
  Ability to Deploy (Right Ventricle): Score 2 | 0
  Ability to Deploy (Right Ventricle): Score 3: number analyzed (Participants) | 8
  Ability to Deploy (Right Ventricle): Score 3 | 0
  Ability to Deploy (Right Ventricle): Score 4: number analyzed (Participants) | 8
  Ability to Deploy (Right Ventricle): Score 4 | 2
  Ability to Deploy (Right Ventricle): Score 5: number analyzed (Participants) | 8
  Ability to Deploy (Right Ventricle): Score 5 | 2
  Ability to Deploy (Right Ventricle): Score 6: number analyzed (Participants) | 8
  Ability to Deploy (Right Ventricle): Score 6 | 4
  Ability to Deploy (Right Ventricle): Score 7: number analyzed (Participants) | 8
  Ability to Deploy (Right Ventricle): Score 7 | 0
  Ability to Maneuver (Left Atrium): Score 1: number analyzed (Participants) | 32
  Ability to Maneuver (Left Atrium): Score 1 | 0
  Ability to Maneuver (Left Atrium): Score 2: number analyzed (Participants) | 32
  Ability to Maneuver (Left Atrium): Score 2 | 1
  Ability to Maneuver (Left Atrium): Score 3: number analyzed (Participants) | 32
  Ability to Maneuver (Left Atrium): Score 3 | 0
  Ability to Maneuver (Left Atrium): Score 4: number analyzed (Participants) | 32
  Ability to Maneuver (Left Atrium): Score 4 | 4
  Ability to Maneuver (Left Atrium): Score 5: number analyzed (Participants) | 32
  Ability to Maneuver (Left Atrium): Score 5 | 8
  Ability to Maneuver (Left Atrium): Score 6: number analyzed (Participants) | 32
  Ability to Maneuver (Left Atrium): Score 6 | 10
  Ability to Maneuver (Left Atrium): Score 7: number analyzed (Participants) | 32
  Ability to Maneuver (Left Atrium): Score 7 | 9
  Ability to Maneuver (Right Atrium): Score 1: number analyzed (Participants) | 17
  Ability to Maneuver (Right Atrium): Score 1 | 0
  Ability to Maneuver (Right Atrium): Score 2: number analyzed (Participants) | 17
  Ability to Maneuver (Right Atrium): Score 2 | 0
  Ability to Maneuver (Right Atrium): Score 3: number analyzed (Participants) | 17
  Ability to Maneuver (Right Atrium): Score 3 | 0
  Ability to Maneuver (Right Atrium): Score 4: number analyzed (Participants) | 17
  Ability to Maneuver (Right Atrium): Score 4 | 1
  Ability to Maneuver (Right Atrium): Score 5: number analyzed (Participants) | 17
  Ability to Maneuver (Right Atrium): Score 5 | 7
  Ability to Maneuver (Right Atrium): Score 6: number analyzed (Participants) | 17
  Ability to Maneuver (Right Atrium): Score 6 | 7
  Ability to Maneuver (Right Atrium): Score 7: number analyzed (Participants) | 17
  Ability to Maneuver (Right Atrium): Score 7 | 2
  Ability to Maneuver (Left Ventricle): Score 1: number analyzed (Participants) | 2
  Ability to Maneuver (Left Ventricle): Score 1 | 0
  Ability to Maneuver (Left Ventricle): Score 2: number analyzed (Participants) | 2
  Ability to Maneuver (Left Ventricle): Score 2 | 0
  Ability to Maneuver (Left Ventricle): Score 3: number analyzed (Participants) | 2
  Ability to Maneuver (Left Ventricle): Score 3 | 0
  Ability to Maneuver (Left Ventricle): Score 4: number analyzed (Participants) | 2
  Ability to Maneuver (Left Ventricle): Score 4 | 1
  Ability to Maneuver (Left Ventricle): Score 5: number analyzed (Participants) | 2
  Ability to Maneuver (Left Ventricle): Score 5 | 0
  Ability to Maneuver (Left Ventricle): Score 6: number analyzed (Participants) | 2
  Ability to Maneuver (Left Ventricle): Score 6 | 0
  Ability to Maneuver (Left Ventricle): Score 7: number analyzed (Participants) | 2
  Ability to Maneuver (Left Ventricle): Score 7 | 1
  Ability to Maneuver (Right Ventricle): Score 1: number analyzed (Participants) | 8
  Ability to Maneuver (Right Ventricle): Score 1 | 0
  Ability to Maneuver (Right Ventricle): Score 2: number analyzed (Participants) | 8
  Ability to Maneuver (Right Ventricle): Score 2 | 0
  Ability to Maneuver (Right Ventricle): Score 3: number analyzed (Participants) | 8
  Ability to Maneuver (Right Ventricle): Score 3 | 0
  Ability to Maneuver (Right Ventricle): Score 4: number analyzed (Participants) | 8
  Ability to Maneuver (Right Ventricle): Score 4 | 2
  Ability to Maneuver (Right Ventricle): Score 5: number analyzed (Participants) | 8
  Ability to Maneuver (Right Ventricle): Score 5 | 2
  Ability to Maneuver (Right Ventricle): Score 6: number analyzed (Participants) | 8
  Ability to Maneuver (Right Ventricle): Score 6 | 3
  Ability to Maneuver (Right Ventricle): Score 7: number analyzed (Participants) | 8
  Ability to Maneuver (Right Ventricle): Score 7 | 1
  Ability to Reach Areas (Left Atrium): Score 1: number analyzed (Participants) | 31
  Ability to Reach Areas (Left Atrium): Score 1 | 0
  Ability to Reach Areas (Left Atrium): Score 2: number analyzed (Participants) | 31
  Ability to Reach Areas (Left Atrium): Score 2 | 1
  Ability to Reach Areas (Left Atrium): Score 3: number analyzed (Participants) | 31
  Ability to Reach Areas (Left Atrium): Score 3 | 0
  Ability to Reach Areas (Left Atrium): Score 4: number analyzed (Participants) | 31
  Ability to Reach Areas (Left Atrium): Score 4 | 4
  Ability to Reach Areas (Left Atrium): Score 5: number analyzed (Participants) | 31
  Ability to Reach Areas (Left Atrium): Score 5 | 7
  Ability to Reach Areas (Left Atrium): Score 6: number analyzed (Participants) | 31
  Ability to Reach Areas (Left Atrium): Score 6 | 11
  Ability to Reach Areas (Left Atrium): Score 7: number analyzed (Participants) | 31
  Ability to Reach Areas (Left Atrium): Score 7 | 8
  Ability to Reach Areas (Right Atrium): Score 1: number analyzed (Participants) | 17
  Ability to Reach Areas (Right Atrium): Score 1 | 0
  Ability to Reach Areas (Right Atrium): Score 2: number analyzed (Participants) | 17
  Ability to Reach Areas (Right Atrium): Score 2 | 0
  Ability to Reach Areas (Right Atrium): Score 3: number analyzed (Participants) | 17
  Ability to Reach Areas (Right Atrium): Score 3 | 0
  Ability to Reach Areas (Right Atrium): Score 4: number analyzed (Participants) | 17
  Ability to Reach Areas (Right Atrium): Score 4 | 2
  Ability to Reach Areas (Right Atrium): Score 5: number analyzed (Participants) | 17
  Ability to Reach Areas (Right Atrium): Score 5 | 5
  Ability to Reach Areas (Right Atrium): Score 6: number analyzed (Participants) | 17
  Ability to Reach Areas (Right Atrium): Score 6 | 8
  Ability to Reach Areas (Right Atrium): Score 7: number analyzed (Participants) | 17
  Ability to Reach Areas (Right Atrium): Score 7 | 2
  Ability to Reach Areas (Left Ventricle): Score 1: number analyzed (Participants) | 2
  Ability to Reach Areas (Left Ventricle): Score 1 | 0
  Ability to Reach Areas (Left Ventricle): Score 2: number analyzed (Participants) | 2
  Ability to Reach Areas (Left Ventricle): Score 2 | 0
  Ability to Reach Areas (Left Ventricle): Score 3: number analyzed (Participants) | 2
  Ability to Reach Areas (Left Ventricle): Score 3 | 0
  Ability to Reach Areas (Left Ventricle): Score 4: number analyzed (Participants) | 2
  Ability to Reach Areas (Left Ventricle): Score 4 | 1
  Ability to Reach Areas (Left Ventricle): Score 5: number analyzed (Participants) | 2
  Ability to Reach Areas (Left Ventricle): Score 5 | 0
  Ability to Reach Areas (Left Ventricle): Score 6: number analyzed (Participants) | 2
  Ability to Reach Areas (Left Ventricle): Score 6 | 0
  Ability to Reach Areas (Left Ventricle): Score 7: number analyzed (Participants) | 2
  Ability to Reach Areas (Left Ventricle): Score 7 | 1
  Ability to Reach Areas (Right Ventricle): Score 1: number analyzed (Participants) | 8
  Ability to Reach Areas (Right Ventricle): Score 1 | 0
  Ability to Reach Areas (Right Ventricle): Score 2: number analyzed (Participants) | 8
  Ability to Reach Areas (Right Ventricle): Score 2 | 0
  Ability to Reach Areas (Right Ventricle): Score 3: number analyzed (Participants) | 8
  Ability to Reach Areas (Right Ventricle): Score 3 | 0
  Ability to Reach Areas (Right Ventricle): Score 4: number analyzed (Participants) | 8
  Ability to Reach Areas (Right Ventricle): Score 4 | 2
  Ability to Reach Areas (Right Ventricle): Score 5: number analyzed (Participants) | 8
  Ability to Reach Areas (Right Ventricle): Score 5 | 3
  Ability to Reach Areas (Right Ventricle): Score 6: number analyzed (Participants) | 8
  Ability to Reach Areas (Right Ventricle): Score 6 | 3
  Ability to Reach Areas (Right Ventricle): Score 7: number analyzed (Participants) | 8
  Ability to Reach Areas (Right Ventricle): Score 7 | 0
  Ability to withdraw (Left Atrium): Score 1: number analyzed (Participants) | 32
  Ability to withdraw (Left Atrium): Score 1 | 0
  Ability to withdraw (Left Atrium): Score 2: number analyzed (Participants) | 32
  Ability to withdraw (Left Atrium): Score 2 | 0
  Ability to withdraw (Left Atrium): Score 3: number analyzed (Participants) | 32
  Ability to withdraw (Left Atrium): Score 3 | 1
  Ability to withdraw (Left Atrium): Score 4: number analyzed (Participants) | 32
  Ability to withdraw (Left Atrium): Score 4 | 6
  Ability to withdraw (Left Atrium): Score 5: number analyzed (Participants) | 32
  Ability to withdraw (Left Atrium): Score 5 | 5
  Ability to withdraw (Left Atrium): Score 6: number analyzed (Participants) | 32
  Ability to withdraw (Left Atrium): Score 6 | 10
  Ability to withdraw (Left Atrium): Score 7: number analyzed (Participants) | 32
  Ability to withdraw (Left Atrium): Score 7 | 10
  Ability to withdraw (Right Atrium): Score 1: number analyzed (Participants) | 19
  Ability to withdraw (Right Atrium): Score 1 | 0
  Ability to withdraw (Right Atrium): Score 2: number analyzed (Participants) | 19
  Ability to withdraw (Right Atrium): Score 2 | 0
  Ability to withdraw (Right Atrium): Score 3: number analyzed (Participants) | 19
  Ability to withdraw (Right Atrium): Score 3 | 0
  Ability to withdraw (Right Atrium): Score 4: number analyzed (Participants) | 19
  Ability to withdraw (Right Atrium): Score 4 | 4
  Ability to withdraw (Right Atrium): Score 5: number analyzed (Participants) | 19
  Ability to withdraw (Right Atrium): Score 5 | 3
  Ability to withdraw (Right Atrium): Score 6: number analyzed (Participants) | 19
  Ability to withdraw (Right Atrium): Score 6 | 9
  Ability to withdraw (Right Atrium): Score 7: number analyzed (Participants) | 19
  Ability to withdraw (Right Atrium): Score 7 | 3
  Ability to withdraw (Left Ventricles): Score 1: number analyzed (Participants) | 2
  Ability to withdraw (Left Ventricles): Score 1 | 0
  Ability to withdraw (Left Ventricles): Score 2: number analyzed (Participants) | 2
  Ability to withdraw (Left Ventricles): Score 2 | 0
  Ability to withdraw (Left Ventricles): Score 3: number analyzed (Participants) | 2
  Ability to withdraw (Left Ventricles): Score 3 | 0
  Ability to withdraw (Left Ventricles): Score 4: number analyzed (Participants) | 2
  Ability to withdraw (Left Ventricles): Score 4 | 0
  Ability to withdraw (Left Ventricles): Score 5: number analyzed (Participants) | 2
  Ability to withdraw (Left Ventricles): Score 5 | 0
  Ability to withdraw (Left Ventricles): Score 6: number analyzed (Participants) | 2
  Ability to withdraw (Left Ventricles): Score 6 | 1
  Ability to withdraw (Left Ventricles): Score 7: number analyzed (Participants) | 2
  Ability to withdraw (Left Ventricles): Score 7 | 1
  Ability to withdraw (Right Ventricles): Score 1: number analyzed (Participants) | 8
  Ability to withdraw (Right Ventricles): Score 1 | 0
  Ability to withdraw (Right Ventricles): Score 2: number analyzed (Participants) | 8
  Ability to withdraw (Right Ventricles): Score 2 | 0
  Ability to withdraw (Right Ventricles): Score 3: number analyzed (Participants) | 8
  Ability to withdraw (Right Ventricles): Score 3 | 0
  Ability to withdraw (Right Ventricles): Score 4: number analyzed (Participants) | 8
  Ability to withdraw (Right Ventricles): Score 4 | 1
  Ability to withdraw (Right Ventricles): Score 5: number analyzed (Participants) | 8
  Ability to withdraw (Right Ventricles): Score 5 | 2
  Ability to withdraw (Right Ventricles): Score 6: number analyzed (Participants) | 8
  Ability to withdraw (Right Ventricles): Score 6 | 4
  Ability to withdraw (Right Ventricles): Score 7: number analyzed (Participants) | 8
  Ability to withdraw (Right Ventricles): Score 7 | 1
  Overall ease of use of the catheter: Score 1 | 0
  Overall ease of use of the catheter: Score 2 | 1
  Overall ease of use of the catheter: Score 3 | 0
  Overall ease of use of the catheter: Score 4 | 6
  Overall ease of use of the catheter: Score 5 | 11
  Overall ease of use of the catheter: Score 6 | 20
  Overall ease of use of the catheter: Score 7 | 2
  Insertion and withdrawal from introducer sheath: Score 1 | 0
  Insertion and withdrawal from introducer sheath: Score 2 | 1
  Insertion and withdrawal from introducer sheath: Score 3 | 0
  Insertion and withdrawal from introducer sheath: Score 4 | 4
  Insertion and withdrawal from introducer sheath: Score 5 | 10
  Insertion and withdrawal from introducer sheath: Score 6 | 13
  Insertion and withdrawal from introducer sheath: Score 7 | 12
  Learning curve: Score 1 | 0
  Learning curve: Score 2 | 1
  Learning curve: Score 3 | 0
  Learning curve: Score 4 | 6
  Learning curve: Score 5 | 12
  Learning curve: Score 6 | 17
  Learning curve: Score 7 | 4

4. Secondary Outcome: Number of Responders for Physician Assessment for Signal Collection and Quality
Description: Number of responders for physician assessment for signal collection and quality (UNIPOLAR signals in atria/ventricles, UNIPOLAR noise encountered, BIPOLAR signals in atria/ventricles, BASELINE noise encountered, and BIPOLAR noise encountered) were reported. A post-procedure survey of 11 questions, each with individual sub-questions were asked. Each question/sub-question was answered by the physician using a Likert scale of 1 to 7 (1=poor and 7=excellent). Responders refers to participants with physician assessment for signal collection and quality.
Time Frame: Up to 29 weeks
Population: The safety analysis set consisted of all enrolled participants who underwent insertion of the study catheter. Here, 'N' (number of participants analyzed) signifies participants evaluated for this outcome measure and 'n' (number analyzed) is defined as participants analyzed for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
Number analyzed (Participants) | 38
Participants
  UNIPOLAR signals in Atria: Score 1: number analyzed (Participants) | 19
  UNIPOLAR signals in Atria: Score 1 | 0
  UNIPOLAR signals in Atria: Score 2: number analyzed (Participants) | 19
  UNIPOLAR signals in Atria: Score 2 | 0
  UNIPOLAR signals in Atria: Score 3: number analyzed (Participants) | 19
  UNIPOLAR signals in Atria: Score 3 | 0
  UNIPOLAR signals in Atria: Score 4: number analyzed (Participants) | 19
  UNIPOLAR signals in Atria: Score 4 | 3
  UNIPOLAR signals in Atria: Score 5: number analyzed (Participants) | 19
  UNIPOLAR signals in Atria: Score 5 | 5
  UNIPOLAR signals in Atria: Score 6: number analyzed (Participants) | 19
  UNIPOLAR signals in Atria: Score 6 | 5
  UNIPOLAR signals in Atria: Score 7: number analyzed (Participants) | 19
  UNIPOLAR signals in Atria: Score 7 | 6
  UNIPOLAR signals in Ventricles: Score 1: number analyzed (Participants) | 9
  UNIPOLAR signals in Ventricles: Score 1 | 0
  UNIPOLAR signals in Ventricles: Score 2: number analyzed (Participants) | 9
  UNIPOLAR signals in Ventricles: Score 2 | 0
  UNIPOLAR signals in Ventricles: Score 3: number analyzed (Participants) | 9
  UNIPOLAR signals in Ventricles: Score 3 | 0
  UNIPOLAR signals in Ventricles: Score 4: number analyzed (Participants) | 9
  UNIPOLAR signals in Ventricles: Score 4 | 2
  UNIPOLAR signals in Ventricles: Score 5: number analyzed (Participants) | 9
  UNIPOLAR signals in Ventricles: Score 5 | 1
  UNIPOLAR signals in Ventricles: Score 6: number analyzed (Participants) | 9
  UNIPOLAR signals in Ventricles: Score 6 | 2
  UNIPOLAR signals in Ventricles: Score 7: number analyzed (Participants) | 9
  UNIPOLAR signals in Ventricles: Score 7 | 4
  UNIPOLAR noise encountered: Score 1: number analyzed (Participants) | 28
  UNIPOLAR noise encountered: Score 1 | 0
  UNIPOLAR noise encountered: Score 2: number analyzed (Participants) | 28
  UNIPOLAR noise encountered: Score 2 | 0
  UNIPOLAR noise encountered: Score 3: number analyzed (Participants) | 28
  UNIPOLAR noise encountered: Score 3 | 0
  UNIPOLAR noise encountered: Score 4: number analyzed (Participants) | 28
  UNIPOLAR noise encountered: Score 4 | 5
  UNIPOLAR noise encountered: Score 5: number analyzed (Participants) | 28
  UNIPOLAR noise encountered: Score 5 | 6
  UNIPOLAR noise encountered: Score 6: number analyzed (Participants) | 28
  UNIPOLAR noise encountered: Score 6 | 11
  UNIPOLAR noise encountered: Score 7: number analyzed (Participants) | 28
  UNIPOLAR noise encountered: Score 7 | 6
  BIPOLAR signals in Atria: Score 1: number analyzed (Participants) | 32
  BIPOLAR signals in Atria: Score 1 | 0
  BIPOLAR signals in Atria: Score 2: number analyzed (Participants) | 32
  BIPOLAR signals in Atria: Score 2 | 0
  BIPOLAR signals in Atria: Score 3: number analyzed (Participants) | 32
  BIPOLAR signals in Atria: Score 3 | 0
  BIPOLAR signals in Atria: Score 4: number analyzed (Participants) | 32
  BIPOLAR signals in Atria: Score 4 | 4
  BIPOLAR signals in Atria: Score 5: number analyzed (Participants) | 32
  BIPOLAR signals in Atria: Score 5 | 6
  BIPOLAR signals in Atria: Score 6: number analyzed (Participants) | 32
  BIPOLAR signals in Atria: Score 6 | 7
  BIPOLAR signals in Atria: Score 7: number analyzed (Participants) | 32
  BIPOLAR signals in Atria: Score 7 | 15
  BIPOLAR signals in Ventricles: Score 1: number analyzed (Participants) | 10
  BIPOLAR signals in Ventricles: Score 1 | 0
  BIPOLAR signals in Ventricles: Score 2: number analyzed (Participants) | 10
  BIPOLAR signals in Ventricles: Score 2 | 0
  BIPOLAR signals in Ventricles: Score 3: number analyzed (Participants) | 10
  BIPOLAR signals in Ventricles: Score 3 | 0
  BIPOLAR signals in Ventricles: Score 4: number analyzed (Participants) | 10
  BIPOLAR signals in Ventricles: Score 4 | 1
  BIPOLAR signals in Ventricles: Score 5: number analyzed (Participants) | 10
  BIPOLAR signals in Ventricles: Score 5 | 0
  BIPOLAR signals in Ventricles: Score 6: number analyzed (Participants) | 10
  BIPOLAR signals in Ventricles: Score 6 | 2
  BIPOLAR signals in Ventricles: Score 7: number analyzed (Participants) | 10
  BIPOLAR signals in Ventricles: Score 7 | 7
  BASELINE noise encountered: Score 1 | 0
  BASELINE noise encountered: Score 2 | 0
  BASELINE noise encountered: Score 3 | 0
  BASELINE noise encountered: Score 4 | 5
  BASELINE noise encountered: Score 5 | 7
  BASELINE noise encountered: Score 6 | 12
  BASELINE noise encountered: Score 7 | 14
  BIPOLAR noise encountered: Score 1 | 0
  BIPOLAR noise encountered: Score 2 | 0
  BIPOLAR noise encountered: Score 3 | 0
  BIPOLAR noise encountered: Score 4 | 5
  BIPOLAR noise encountered: Score 5 | 9
  BIPOLAR noise encountered: Score 6 | 9
  BIPOLAR noise encountered: Score 7 | 15

5. Secondary Outcome: Number of Responders for Physician Assessment for Pacing
Description: Number of responders for physician assessment for pacing (high output stimulation pacing and local pacing capture) were reported. A post-procedure survey of 11 questions, each with individual sub-questions were asked. Each question/sub-question was answered by the physician using a Likert scale of 1 to 7 (1=poor and 7=excellent). Responders refers to participants with physician assessment for pacing.
Time Frame: Up to 29 weeks
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
Number analyzed (Participants) | 23
Participants
  High output stimulation pacing: Score 1: number analyzed (Participants) | 5
  High output stimulation pacing: Score 1 | 0
  High output stimulation pacing: Score 2: number analyzed (Participants) | 5
  High output stimulation pacing: Score 2 | 0
  High output stimulation pacing: Score 3: number analyzed (Participants) | 5
  High output stimulation pacing: Score 3 | 0
  High output stimulation pacing: Score 4: number analyzed (Participants) | 5
  High output stimulation pacing: Score 4 | 1
  High output stimulation pacing: Score 5: number analyzed (Participants) | 5
  High output stimulation pacing: Score 5 | 1
  High output stimulation pacing: Score 6: number analyzed (Participants) | 5
  High output stimulation pacing: Score 6 | 1
  High output stimulation pacing: Score 7: number analyzed (Participants) | 5
  High output stimulation pacing: Score 7 | 2
  Local pacing capture: Score 1 | 0
  Local pacing capture: Score 2 | 1
  Local pacing capture: Score 3 | 2
  Local pacing capture: Score 4 | 4
  Local pacing capture: Score 5 | 7
  Local pacing capture: Score 6 | 4
  Local pacing capture: Score 7 | 5

6. Secondary Outcome: Number of Responders for Physician Assessment for Catheter Design
Description: Number of responders for physician assessment for catheter design were reported. A post-procedure survey of 11 questions, each with individual sub-questions were asked. Each question/sub-question was answered by the physician using a Likert scale of 1 to 7 (1=poor and 7=excellent). Responders refers to participants with physician assessment for catheter design.
Time Frame: Up to 29 weeks
Population: The safety analysis set consisted of all enrolled participants who underwent insertion of the study catheter.
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
Number analyzed (Participants) | 40
Participants
  Ability to achieve electrode contact with cardiac tissue: Score 1 | 0
  Ability to achieve electrode contact with cardiac tissue: Score 2 | 1
  Ability to achieve electrode contact with cardiac tissue: Score 3 | 0
  Ability to achieve electrode contact with cardiac tissue: Score 4 | 4
  Ability to achieve electrode contact with cardiac tissue: Score 5 | 11
  Ability to achieve electrode contact with cardiac tissue: Score 6 | 22
  Ability to achieve electrode contact with cardiac tissue: Score 7 | 2
  Electrodes spacing: Score 1 | 0
  Electrodes spacing: Score 2 | 0
  Electrodes spacing: Score 3 | 0
  Electrodes spacing: Score 4 | 4
  Electrodes spacing: Score 5 | 10
  Electrodes spacing: Score 6 | 13
  Electrodes spacing: Score 7 | 13
  Electrode array coverage: Score 1 | 0
  Electrode array coverage: Score 2 | 0
  Electrode array coverage: Score 3 | 0
  Electrode array coverage: Score 4 | 4
  Electrode array coverage: Score 5 | 10
  Electrode array coverage: Score 6 | 18
  Electrode array coverage: Score 7 | 8

7. Secondary Outcome: Number of Responders for Physician Assessment for Workflow
Description: Number of responders for physician assessment for workflow were reported. A post-procedure survey of 11 questions, each with individual sub-questions were asked. Each question/sub-question was answered by the physician using a Likert scale of 1 to 7 (1=poor and 7=excellent). Responders refers to participants with physician assessment for workflow.
Time Frame: Up to 29 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
Number analyzed (Participants) | 40
Participants
  Ability to reduce fluoroscopy: Score 1: number analyzed (Participants) | 38
  Ability to reduce fluoroscopy: Score 1 | 0
  Ability to reduce fluoroscopy: Score 2: number analyzed (Participants) | 38
  Ability to reduce fluoroscopy: Score 2 | 1
  Ability to reduce fluoroscopy: Score 3: number analyzed (Participants) | 38
  Ability to reduce fluoroscopy: Score 3 | 4
  Ability to reduce fluoroscopy: Score 4: number analyzed (Participants) | 38
  Ability to reduce fluoroscopy: Score 4 | 5
  Ability to reduce fluoroscopy: Score 5: number analyzed (Participants) | 38
  Ability to reduce fluoroscopy: Score 5 | 14
  Ability to reduce fluoroscopy: Score 6: number analyzed (Participants) | 38
  Ability to reduce fluoroscopy: Score 6 | 4
  Ability to reduce fluoroscopy: Score 7: number analyzed (Participants) | 38
  Ability to reduce fluoroscopy: Score 7 | 10
  Time for pre-procedure mapping: Score 1 | 0
  Time for pre-procedure mapping: Score 2 | 1
  Time for pre-procedure mapping: Score 3 | 0
  Time for pre-procedure mapping: Score 4 | 4
  Time for pre-procedure mapping: Score 5 | 14
  Time for pre-procedure mapping: Score 6 | 19
  Time for pre-procedure mapping: Score 7 | 2
  Time for post-procedure mapping after standard of care ablation: Score 1: number analyzed (Participants) | 36
  Time for post-procedure mapping after standard of care ablation: Score 1 | 0
  Time for post-procedure mapping after standard of care ablation: Score 2: number analyzed (Participants) | 36
  Time for post-procedure mapping after standard of care ablation: Score 2 | 1
  Time for post-procedure mapping after standard of care ablation: Score 3: number analyzed (Participants) | 36
  Time for post-procedure mapping after standard of care ablation: Score 3 | 0
  Time for post-procedure mapping after standard of care ablation: Score 4: number analyzed (Participants) | 36
  Time for post-procedure mapping after standard of care ablation: Score 4 | 4
  Time for post-procedure mapping after standard of care ablation: Score 5: number analyzed (Participants) | 36
  Time for post-procedure mapping after standard of care ablation: Score 5 | 8
  Time for post-procedure mapping after standard of care ablation: Score 6: number analyzed (Participants) | 36
  Time for post-procedure mapping after standard of care ablation: Score 6 | 11
  Time for post-procedure mapping after standard of care ablation: Score 7: number analyzed (Participants) | 36
  Time for post-procedure mapping after standard of care ablation: Score 7 | 12
  Ability to identify targets: Score 1: number analyzed (Participants) | 29
  Ability to identify targets: Score 1 | 0
  Ability to identify targets: Score 2: number analyzed (Participants) | 29
  Ability to identify targets: Score 2 | 0
  Ability to identify targets: Score 3: number analyzed (Participants) | 29
  Ability to identify targets: Score 3 | 0
  Ability to identify targets: Score 4: number analyzed (Participants) | 29
  Ability to identify targets: Score 4 | 4
  Ability to identify targets: Score 5: number analyzed (Participants) | 29
  Ability to identify targets: Score 5 | 11
  Ability to identify targets: Score 6: number analyzed (Participants) | 29
  Ability to identify targets: Score 6 | 9
  Ability to identify targets: Score 7: number analyzed (Participants) | 29
  Ability to identify targets: Score 7 | 5

8. Secondary Outcome: Number of Responders for Physician Assessment for Catheter Visualization
Description: Number of responders for physician assessment for catheter visualization were reported. A post-procedure survey of 11 questions, each with individual sub-questions were asked. Each question/sub-question was answered by the physician using a Likert scale of 1 to 7 (1=poor and 7=excellent). Responders refers to participants with physician assessment for catheter visualization.
Time Frame: Up to 29 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
Number analyzed (Participants) | 40
Participants
  Visualization under fluoroscopy: Score 1: number analyzed (Participants) | 38
  Visualization under fluoroscopy: Score 1 | 0
  Visualization under fluoroscopy: Score 2: number analyzed (Participants) | 38
  Visualization under fluoroscopy: Score 2 | 2
  Visualization under fluoroscopy: Score 3: number analyzed (Participants) | 38
  Visualization under fluoroscopy: Score 3 | 0
  Visualization under fluoroscopy: Score 4: number analyzed (Participants) | 38
  Visualization under fluoroscopy: Score 4 | 5
  Visualization under fluoroscopy: Score 5: number analyzed (Participants) | 38
  Visualization under fluoroscopy: Score 5 | 10
  Visualization under fluoroscopy: Score 6: number analyzed (Participants) | 38
  Visualization under fluoroscopy: Score 6 | 18
  Visualization under fluoroscopy: Score 7: number analyzed (Participants) | 38
  Visualization under fluoroscopy: Score 7 | 3
  Visualization in CARTO 3: Score 1 | 0
  Visualization in CARTO 3: Score 2 | 0
  Visualization in CARTO 3: Score 3 | 4
  Visualization in CARTO 3: Score 4 | 6
  Visualization in CARTO 3: Score 5 | 9
  Visualization in CARTO 3: Score 6 | 9
  Visualization in CARTO 3: Score 7 | 12

9. Secondary Outcome: Number of Responders for Physician Assessment for Catheters Interactions
Description: Number of responders for physician assessment for catheters interactions were reported. A post-procedure survey of 11 questions, each with individual sub-questions were asked. Each question/sub-question was answered by the physician using a Likert scale of 1 to 7 (1=poor and 7=excellent). Responders refers to participants with physician assessment for catheters interactions.
Time Frame: Up to 29 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
Number analyzed (Participants) | 40
Participants
  CARTO 3 System: Score 1 | 1
  CARTO 3 System: Score 2 | 0
  CARTO 3 System: Score 3 | 2
  CARTO 3 System: Score 4 | 7
  CARTO 3 System: Score 5 | 10
  CARTO 3 System: Score 6 | 16
  CARTO 3 System: Score 7 | 4
  Electrophysiology (EP) Lab recording equipment: Score 1 | 1
  EP Lab recording equipment: Score 2 | 0
  EP Lab recording equipment: Score 3 | 2
  EP Lab recording equipment: Score 4 | 6
  EP Lab recording equipment: Score 5 | 16
  EP Lab recording equipment: Score 6 | 11
  EP Lab recording equipment: Score 7 | 4
  Pacing equipment: Score 1: number analyzed (Participants) | 27
  Pacing equipment: Score 1 | 0
  Pacing equipment: Score 2: number analyzed (Participants) | 27
  Pacing equipment: Score 2 | 0
  Pacing equipment: Score 3: number analyzed (Participants) | 27
  Pacing equipment: Score 3 | 0
  Pacing equipment: Score 4: number analyzed (Participants) | 27
  Pacing equipment: Score 4 | 4
  Pacing equipment: Score 5: number analyzed (Participants) | 27
  Pacing equipment: Score 5 | 12
  Pacing equipment: Score 6: number analyzed (Participants) | 27
  Pacing equipment: Score 6 | 3
  Pacing equipment: Score 7: number analyzed (Participants) | 27
  Pacing equipment: Score 7 | 8
  Introducer tool on catheter: Score 1 | 1
  Introducer tool on catheter: Score 2 | 1
  Introducer tool on catheter: Score 3 | 0
  Introducer tool on catheter: Score 4 | 5
  Introducer tool on catheter: Score 5 | 8
  Introducer tool on catheter: Score 6 | 13
  Introducer tool on catheter: Score 7 | 12
  Sheath: Score 1 | 1
  Sheath: Score 2 | 1
  Sheath: Score 3 | 0
  Sheath: Score 4 | 5
  Sheath: Score 5 | 9
  Sheath: Score 6 | 12
  Sheath: Score 7 | 12
  Irrigation bag and tubing: Score 1 | 1
  Irrigation bag and tubing: Score 2 | 0
  Irrigation bag and tubing: Score 3 | 0
  Irrigation bag and tubing: Score 4 | 6
  Irrigation bag and tubing: Score 5 | 9
  Irrigation bag and tubing: Score 6 | 12
  Irrigation bag and tubing: Score 7 | 12
  Implantable cardioverter-defibrillators (ICD) or other implantable devices: Score 1: number analyzed (Participants) | 1
  Implantable cardioverter-defibrillators (ICD) or other implantable devices: Score 1 | 0
  ICD or other implantable devices: Score 2: number analyzed (Participants) | 1
  ICD or other implantable devices: Score 2 | 0
  ICD or other implantable devices: Score 3: number analyzed (Participants) | 1
  ICD or other implantable devices: Score 3 | 0
  ICD or other implantable devices: Score 4: number analyzed (Participants) | 1
  ICD or other implantable devices: Score 4 | 0
  ICD or other implantable devices: Score 5: number analyzed (Participants) | 1
  ICD or other implantable devices: Score 5 | 0
  ICD or other implantable devices: Score 6: number analyzed (Participants) | 1
  ICD or other implantable devices: Score 6 | 1
  ICD or other implantable devices: Score 7: number analyzed (Participants) | 1
  ICD or other implantable devices: Score 7 | 0

10. Secondary Outcome: Number of Responders for Physician Assessment for Arrhythmogenicity
Description: Number of responders for physician assessment for arrhythmogenicity were reported. A post-procedure survey of 11 questions, each with individual sub-questions were asked. Each question/sub-question was answered by the physician using a Likert scale of 1 to 7 (1=poor and 7=excellent). Responders refers to participants with physician assessment for arrhythmogenicity.
Time Frame: Up to 29 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
Number analyzed (Participants) | 40
Participants
  Compared to the PENTARAY catheter: Score 1 | 0
  Compared to the PENTARAY catheter: Score 2 | 0
  Compared to the PENTARAY catheter: Score 3 | 1
  Compared to the PENTARAY catheter: Score 4 | 1
  Compared to the PENTARAY catheter: Score 5 | 10
  Compared to the PENTARAY catheter: Score 6 | 20
  Compared to the PENTARAY catheter: Score 7 | 8
  Compared to other competitive multielectrode catheters: Score 1: number analyzed (Participants) | 29
  Compared to other competitive multielectrode catheters: Score 1 | 0
  Compared to other competitive multielectrode catheters: Score 2: number analyzed (Participants) | 29
  Compared to other competitive multielectrode catheters: Score 2 | 0
  Compared to other competitive multielectrode catheters: Score 3: number analyzed (Participants) | 29
  Compared to other competitive multielectrode catheters: Score 3 | 1
  Compared to other competitive multielectrode catheters: Score 4: number analyzed (Participants) | 29
  Compared to other competitive multielectrode catheters: Score 4 | 5
  Compared to other competitive multielectrode catheters: Score 5: number analyzed (Participants) | 29
  Compared to other competitive multielectrode catheters: Score 5 | 7
  Compared to other competitive multielectrode catheters: Score 6: number analyzed (Participants) | 29
  Compared to other competitive multielectrode catheters: Score 6 | 12
  Compared to other competitive multielectrode catheters: Score 7: number analyzed (Participants) | 29
  Compared to other competitive multielectrode catheters: Score 7 | 4

11. Secondary Outcome: Number of Responders for Physician Assessment for Design and Coverage for Confirming Pulmonary Vein Isolation (PVI)
Description: Number of responders for physician assessment for design and coverage for confirming PVI were reported. A post-procedure survey of 11 questions, each with individual sub-questions were asked. Each question/sub-question was answered by the physician using a Likert scale of 1 to 7 (1=poor and 7=excellent). Responders refers to participants with physician assessment for design and coverage for confirming PVI.
Time Frame: Up to 29 weeks
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
Number analyzed (Participants) | 30
Participants
  Compared to the PENTARAY catheter: Score 1 | 0
  Compared to the PENTARAY catheter: Score 2 | 0
  Compared to the PENTARAY catheter: Score 3 | 1
  Compared to the PENTARAY catheter: Score 4 | 1
  Compared to the PENTARAY catheter: Score 5 | 8
  Compared to the PENTARAY catheter: Score 6 | 12
  Compared to the PENTARAY catheter: Score 7 | 8
  Compared to other competitive multielectrode catheters: Score 1: number analyzed (Participants) | 21
  Compared to other competitive multielectrode catheters: Score 1 | 0
  Compared to other competitive multielectrode catheters: Score 2: number analyzed (Participants) | 21
  Compared to other competitive multielectrode catheters: Score 2 | 0
  Compared to other competitive multielectrode catheters: Score 3: number analyzed (Participants) | 21
  Compared to other competitive multielectrode catheters: Score 3 | 1
  Compared to other competitive multielectrode catheters: Score 4: number analyzed (Participants) | 21
  Compared to other competitive multielectrode catheters: Score 4 | 1
  Compared to other competitive multielectrode catheters: Score 5: number analyzed (Participants) | 21
  Compared to other competitive multielectrode catheters: Score 5 | 10
  Compared to other competitive multielectrode catheters: Score 6: number analyzed (Participants) | 21
  Compared to other competitive multielectrode catheters: Score 6 | 6
  Compared to other competitive multielectrode catheters: Score 7: number analyzed (Participants) | 21
  Compared to other competitive multielectrode catheters: Score 7 | 3

12. Secondary Outcome: Number of Responders for Physician Assessment for Ability to Characterize the Tissue
Description: Number of responders for physician assessment for ability to characterize the tissue were reported. A post-procedure survey of 11 questions, each with individual sub-questions were asked. Each question/sub-question was answered by the physician using a Likert scale of 1 to 7 (1=poor and 7=excellent). Responders refers to participants with physician assessment for ability to characterize the tissue.
Time Frame: Up to 29 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
Number analyzed (Participants) | 40
Participants
  Compared to the PENTARAY catheter: Score 1 | 0
  Compared to the PENTARAY catheter: Score 2 | 0
  Compared to the PENTARAY catheter: Score 3 | 1
  Compared to the PENTARAY catheter: Score 4 | 5
  Compared to the PENTARAY catheter: Score 5 | 10
  Compared to the PENTARAY catheter: Score 6 | 17
  Compared to the PENTARAY catheter: Score 7 | 7
  Compared to other competitive multielectrode catheters: Score 1: number analyzed (Participants) | 28
  Compared to other competitive multielectrode catheters: Score 1 | 0
  Compared to other competitive multielectrode catheters: Score 2: number analyzed (Participants) | 28
  Compared to other competitive multielectrode catheters: Score 2 | 0
  Compared to other competitive multielectrode catheters: Score 3: number analyzed (Participants) | 28
  Compared to other competitive multielectrode catheters: Score 3 | 0
  Compared to other competitive multielectrode catheters: Score 4: number analyzed (Participants) | 28
  Compared to other competitive multielectrode catheters: Score 4 | 8
  Compared to other competitive multielectrode catheters: Score 5: number analyzed (Participants) | 28
  Compared to other competitive multielectrode catheters: Score 5 | 9
  Compared to other competitive multielectrode catheters: Score 6: number analyzed (Participants) | 28
  Compared to other competitive multielectrode catheters: Score 6 | 10
  Compared to other competitive multielectrode catheters: Score 7: number analyzed (Participants) | 28
  Compared to other competitive multielectrode catheters: Score 7 | 1

13. Secondary Outcome: Number of Responders for Physician Assessment for Ability to Identify Arrhythmia Circuit or Source Correctly
Description: Number of responders for physician assessment for ability to identify arrhythmia circuit or source correctly were reported. A post-procedure survey of 11 questions, each with individual sub-questions were asked. Each question/sub-question was answered by the physician using a Likert scale of 1 to 7 (1=poor and 7=excellent). Responders refers to participants with physician assessment for ability to identify arrhythmia circuit or source correctly.
Time Frame: Up to 29 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
Number analyzed (Participants) | 40
Participants
  Compared to the PENTARAY catheter: Score 1 | 0
  Compared to the PENTARAY catheter: Score 2 | 1
  Compared to the PENTARAY catheter: Score 3 | 0
  Compared to the PENTARAY catheter: Score 4 | 3
  Compared to the PENTARAY catheter: Score 5 | 14
  Compared to the PENTARAY catheter: Score 6 | 18
  Compared to the PENTARAY catheter: Score 7 | 4
  Compared to other competitive multielectrode catheters: Score 1: number analyzed (Participants) | 28
  Compared to other competitive multielectrode catheters: Score 1 | 0
  Compared to other competitive multielectrode catheters: Score 2: number analyzed (Participants) | 28
  Compared to other competitive multielectrode catheters: Score 2 | 0
  Compared to other competitive multielectrode catheters: Score 3: number analyzed (Participants) | 28
  Compared to other competitive multielectrode catheters: Score 3 | 1
  Compared to other competitive multielectrode catheters: Score 4: number analyzed (Participants) | 28
  Compared to other competitive multielectrode catheters: Score 4 | 5
  Compared to other competitive multielectrode catheters: Score 5: number analyzed (Participants) | 28
  Compared to other competitive multielectrode catheters: Score 5 | 14
  Compared to other competitive multielectrode catheters: Score 6: number analyzed (Participants) | 28
  Compared to other competitive multielectrode catheters: Score 6 | 7
  Compared to other competitive multielectrode catheters: Score 7: number analyzed (Participants) | 28
  Compared to other competitive multielectrode catheters: Score 7 | 1

14. Secondary Outcome: Number of Participants With SAEs Excluding Investigational Catheter Related Within 7 Days of Index Procedure
Description: Number of participants with SAEs excluding investigational catheter related within 7 days of index procedure were reported. An AE is any untoward medical occurrence in a participant whether or not related to the investigational device. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to 7 days of index procedure on Day 1
Population: The safety analysis set consisted of all enrolled participants who underwent insertion of the study catheter.
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
Number analyzed (Participants) | 40
Participants | 3

15. Secondary Outcome: Number of Participants With Non-serious Adverse Events Within 7 Days of Index Procedure Related to the Investigational Catheter
Description: Number of participants with non-serious AEs within 7 days of index procedure related to the investigational catheter were reported. An AE is any untoward medical occurrence in a participant whether or not related to the investigational device.
Time Frame: Up to 7 days of index procedure on Day 1
Population: The safety analysis set consisted of all enrolled participants who underwent insertion of the study catheter.
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
Number analyzed (Participants) | 40
Participants | 1

ADVERSE EVENTS:
Time Frame: From screening up to 29 weeks
Description: The safety analysis set consisted of all enrolled participants who underwent insertion of the study catheter.
Arm/Group | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter)
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 4/40
Other Adverse Events (participants affected / at risk) | 1/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter) (N=40)
Atrioventricular block (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Transient complete atrioventricular block (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multi-electrode Electrocardiogram (ECG) Mapping Catheter (Investigational Catheter) (N=40)
Transient right bundle branch block (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study results/conclusions were based on descriptive analysis due to small sample size. Identification of arrhythmia's mechanism was based on common types of arrhythmias, not for all arrhythmias. Comparisons of globe-shaped design with other multi-electrode catheters could only be performed based on physician feedback in the post-procedure survey. Although CARTO system being the latest version, no specific features were developed to maximize the use of catheter's globe-shape design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications and/or presentation of clinical investigation results will be coordinated and governed between Biosense Webster, Inc., the clinical investigation author(s) and if applicable local law. Authorship will be determined prior to development of any manuscript.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT05373862/Prot_SAP_000.pdf